CLINICAL TRIAL: NCT04152967
Title: New Designed ePTFE Valved Conduits for Surgical Reconstruction of Right-ventricular Outflow Tract: A Multi-centre Clinical Research
Brief Title: New Designed ePTFE Valved Conduits for Surgical Reconstruction of Right-ventricular Outflow Tract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JB-PTFE
Record Dates: First submitted 2019-10-30; First posted 2019-11-06 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Right Ventricular Outflow Tract Absent; Congenital Heart Disease; Pulmonary Valve Disorders
Keywords: PTFE valved conduit; right ventricular outflow tract
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Patients involved in this research should meet the requirement that they need valved conduits to reconstruct right ventricular outflow tract, first time operation and reoperation to change the decayed conduit included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new-designed PTFE valved conduit (Experimental): In this group, new-designed PTFE valved conduits will be applied for patients.
  Interventions: Device: new-designed PTFE valved conduits
- Bovine jugular valved conduit (Active Comparator): In this group, bovine jugular vein valved conduits will be applied for patients.
  Interventions: Device: Bovine jugular vein valved conduits

INTERVENTIONS:
Device: new-designed PTFE valved conduits — In this prospective comparative research, all patients will be divided into two groups randomly with 100 patients in each group. One group will use the new-designed PTFE valved conduits and another one will implant the bovine jugular vein valved conduits.
  Arms: new-designed PTFE valved conduit
Device: Bovine jugular vein valved conduits — In this prospective comparative research, all patients will be divided into two groups randomly with 100 patients in each group. One group will use the new-designed PTFE valved conduits and another one will implant the bovine jugular vein valved conduits.
  Arms: Bovine jugular valved conduit

SUMMARY:
Valved conduits used for the reconstruction of right-ventricular outflow tract are applied in the surgical repair of complex congenital heart disease(CHD) such as pulmonary atresia(PA), truncus arteriosus, severe tetralogy of Fallot(TOF) for their significant roles in reducing pulmonary valve regurgitation and preserving right ventricle function. With a rising cases of complex CHD and patients with pulmonary valve regurgitation in TOF repair, a further demand is underway for valved conduits. Meanwhile, common biological valved conduits applied in foreign countries are not approved in China yet, with high failure and reintervention, reducing the long-term survival. Our team manufactured a novel valved conduit with 0.1mm expanded polytetrafluoroethylene and gore-tex conduit. This ePTFE valved conduit played a satisfying role in anti-regurgitation and failure rate through in vitro fluid test and animal experiments. Besides, our team manufactured templates for the conduit and also simplified the suturing process so that the repeatability of suturing valved had been risen. Until now, over 70 cases have been implanted with this ePTFE valved conduit with positive early and mid-term follow-up results.

Despite the progress which have been made, there still remain some problems to solve. First, systematic prospective randomized comparative study will be performed. Second, this is just a single-center study. Third, these patients should have longer follow-up time to evaluate the ePTFE conduit long-term effect. Finally, imaging data are blank for evaluating the function of the conduit and right ventricle. In this prospective comparative research, the new designed ePTFE valved conduit and bovine jugular vein valved conduits are conducted as a randomized controlled trail. Cardiac magnetic resonance imaging is used to precisely evaluate the anti-regurgitation effect of the valved conduit and the right ventricle function. Investigators can further access the application of this newly designed ePTFE valved conduit. Investigators aim to provide a self-manufactured, low failure rate valved conduit.

DETAILED DESCRIPTION:
Valved conduits used for the reconstruction of right-ventricular outflow tract are applied in the surgical repair of complex congenital heart disease(CHD) such as pulmonary atresia(PA), truncus arteriosus, severe tetralogy of Fallot(TOF) for their significant roles in reducing pulmonary valve regurgitation and preserving right ventricle function. With a rising cases of complex CHD and patients after surgical repair of TOF with pulmonary valve regurgitation, a progressive need is underway for valved conduits. Meanwhile, biological valved conduits used in foreign countries are lacked in China, with the disadvantage that a high failure rate of biological conduits increasing the chances of reoperation which greatly reduce the long-term survival rate. Thus, a new, low failure rate valved conduit with effective performance is urgently needed.

Our team manufactured a new valved conduit with 0.1mm expanded polytetrafluoroethylene and blood vessels. This valved conduit exhibited a fine anti-regurgitation effect and a relatively low failure rate through in vitro fluid test and animal model. Besides, our team manufactured templates for the conduit and also simplified the suturing process so that the repeatability of suturing valved had been risen. Our team have already applied a patent for inventing and a utility model patent for this technique. Several papers have also been published.

Till now, over 70 cases have been involved with this valved conduit with positive early and mid-term follow-up results. Our team have promoted this technique to several heart center such as Zhongshan Hospital affiliated to Fudan University, Shanghai Children's Medical Center and Nanjing Children's Hospital and all department have achieved satisfactory effects.

Despite the progress which have been made, there are still problems remained to be solved to prove the superiority of valved conduits. First, systematic prospective comparative study is required. Second, 70 cases are not enough and currently this is just a single-center study. Third, follow-up time is too short to evaluate the long-term effect. Last but not least, imaging data are blank for evaluating the function of the conduit and right ventricle.

In this prospective comparative research, the new designed PTFE valved conduit and bovine jugular vein valved conduits are conducted as a randomized controlled trail. Cardiac magnetic resonance imaging is used to precisely evaluate the anti-regurgitation effect of the valved conduit and the right ventricle function. Investigators can further access the application of this newly designed PTFE valved conduit. Investigators aim to provide a self-manufactured, low failure rate valved conduit.

Method

1. Patients involved in this research should meet the requirement that they need valved conduits to reconstruct right ventricular outflow tract, first time operation and reoperation to change the fail conduit included. Our team expect 200 patients to meet the requirement.
2. In this prospective comparative research, all patients will be divided into two groups randomly with 100 patients in each group. One group will use the new-designed PTFE valved conduits and another one will implant the bovine jugular vein valved conduits.
3. All patients will receive standard cardiopulmonary bypass through a mid-sternum incision and new-designed PTFE valved conduits or bovine jugular vein valved conduits will be implanted.
4. Pre-operation, operation and post-operation materials will be collected. Besides, every one month, three months, six months, twelve months and twenty-for months after surgery, echocardiography and electrocardiogram will be conducted on each patient. 12 months and 24 months after the surgery, our team will arrange MRI test with the patient on telephone.
5. Assessment:

i. Echocardiography: regurgitation of the valve in the conduits, the position of the regurgitation, the length of matched valve margin, volume of right ventricle, velocity of blood flow through pulmonary valve and pressure gradient will be monitored.

ii. Electrocardiography: arrhythmia and the width of 'QRS' wave. iii. MRI: regurgitation index of valved conduit, RVEDVI, RVESVI, McGoon index, NAKATA index, d survival rate, free from stenosis rate, free from reintervention rate, free from endocarditis rate.

f) MRI test: Using a Siemens Avanto 1.5T MRI spectrometer with a retrospective gated rate coding sequence to conduct the examination. Scanning parameters are set at view 400 mm, TR27 ms, TE 3.2 ms, matrix 240 x 256, layer thickness 5 mm, flip angle 30 degrees. Patients will breath calmly and apply the iPAT (parallel acquisition) technology to reduce imaging time and artifacts. The average examination time will be 20 to 30 minutes.

i. Measurements of valve regurgitation of the conduit: Take the sagittal long axis section of the right ventricular outflow tract and locate it at the level of the valve, and set the flow rate at 200 cm/s to produce a phase contrast sequence diagram. The valve section is circled where white represents the forward blood flow signal and black represents the reflux blood flow signal. The pulmonary flow velocity-time curve is generated by Argus software and calculate the pulmonary artery forward blood flow (FFV) and reverse blood flow (BFV). 2 measurements were taken and averaged. The regurgitation index will be calculated according to the formula BFV/FFV × 100%.

ii. Measurements of right ventricle function: Using a Siemens Avanto 1.5T MRI spectrometer with the Truefisp or flash flair. Scanning parameters are set at view 400 mm, TR2.2 ms, TE 1.5 ms, matrix 128 x 256, layer thickness 5 mm, flip angle 45 degrees. Patients will breath calmly and apply the iPAT (parallel acquisition) technology to reduce imaging time and artifacts. In the short-axis view of the ventricle, the contours of each layer's endocardium at the end of diastolic and end-systolic phases of the right ventricle will be traced, and RVEDV, RVESV, and RVEF will be generated by Argus software.

g) Echocardiography examination: Images will be collected and stored using the PhiliPsIE33 color ultrasound system. The parameters including RVEDV, RVESV, and RVEF will be measured on the machine using QLAB 4.0 software.

Manufacture the new designed conduit: First, turn the inner surface of the conduit to the outside of the conduit and then use template A to draw the stitching positions(three "T" lines and three midpoints). After that, apply template B to draw on 0.1mm PTFE patch and cut into three connected "U" shapes, surrounding the conduit. Suture the patch to the conduit before restoring the conduit to normal. The valve is formed at the boundary. (0.1mm PTFE patch and conduits have been used clinically, provided by Gore)

Reconstruction of the right ventricle outflow tract:

All patients will be divided randomly into two groups. One will implant the new-designed PTFE valved conduits and another one will implant the bovine jugular vein valved conduits.

A mid-sternum incision will be applied for each patient and standard cardiopulmonary bypass will be constructed. Cardiac malformation will be repaired under cardiac arrest. The new-designed PTFE conduit or bovine jugular conduit will be used to connect the right ventricle and pulmonary artery. The distal end of the valved conduit is cut into a bevel surface, and the end of the conduit is merged with the pulmonary artery for end-to-end anastomosis, so that the valve can get closer to the pulmonary artery which will reduce the possibility of valve regurgitation due to blood flow filling pulmonary artery. After the anastomosis, the aorta clutch will be removed, and the heartbeat will recover. The next step is to start the anastomosis of the proximal end and right ventricular. The posterior wall of the anastomosis is sutured directly, and the anterior wall is expanded with autologous pericardium to avoid the narrowing of the proximal anastomosis.

Postoperative anticoagulation: Heparin will be administered intravenously 5~15u/kg/h 4 to 6 hours after surgery if without active hemorrhage. After that, oral anticoagulation with warfarin will be used for 6 months, and the INR should be maintained at 1.5~2.5. 6 months later aspirin will replace warfarin with 3 ~ 5mg / kg / time, once a day, until 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients need valved conduits to reconstruct right ventricular outflow tract, first time operation and reoperation to change the fail conduit included

Exclusion Criteria:

* patients with infective endocarditis before surgery;
* systemic immune disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Regurgitatioin Index of Valve Conduit by Cardiac MRI | twenty-four months after surgery
  Detect pulmonary artery forward blood flow (FFV) and reverse blood flow (BFV) by MRI. PR Index=BFV/FFV × 100%.

SECONDARY OUTCOMES:
arrhythmia using electrocardiogram | three months after surgery
  atril arrhythmia and/or ventricular arrhythmia
arrhythmia using electrocardiogram | six months after surgery
  atril arrhythmia and/or ventricular arrhythmia
arrhythmia using electrocardiogram | twelve months after surgery
  atril arrhythmia and/or ventricular arrhythmia
arrhythmia using electrocardiogram | twenty-four months after surgery
  atril arrhythmia and/or ventricular arrhythmia
pressure gradient across the valve by echocardiography | twenty-four months after surgery
  pressure gradient across the valve detected by dopplor echocardiography
pressure gradient across the valve by echocardiography | one month after surgery
  pressure gradient across the valve detected by dopplor echocardiography
pressure gradient across the valve by echocardiography | three months after surgery
  pressure gradient across the valve detected by dopplor echocardiography
pressure gradient over the valve using Echocardiography | six months after surgery
  pressure gradient across the valve detected by dopplor echocardiography
pressure gradient across the valve by echocardiography | twelve months after surgery
  pressure gradient across the valve detected by dopplor echocardiography
right ventricular end-diastolic volume index by cardiac MRI | twelve months after surgery
  right ventricular end-diastolic volume index detected by MRI
right ventricular end-diastolic volume index by cardiac MRI | twenty-four months after surgery
  right ventricular end-diastolic volume index detected by MRI
McGoon index by Cardiac MRI | twenty-four months after surgery
  McGoon index
McGoon index by Cardiac MRI | twelve months after surgery
  McGoon index
NAKATA index by Cardiac MRI | twelve months after surgery
  NAKATA index
NAKATA index by Cardiac MRI | twenty-four months after surgery
  NAKATA index

CONTACTS AND LOCATIONS:
Overall Officials: Bing Jia, PhD, Study Chair — Children's Hospital of Fudan University
Locations (3):
- China (3):
  - Children's Hospital of Fudan University, Shanghai
  - Shanghai Children's medical center, Shanghai
  - Shanghai zhongshan hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No
Under discussion.

REFERENCES:
- [Background] Hoashi T, Iwasa T, Kagisaki K, Shimada M, Kurosaki K, Shiraishi I, Ichikawa H. Long-term respiratory outcomes after primary total correction for tetralogy of Fallot and absent pulmonary valve in patient with respiratory symptoms. Congenit Heart Dis. 2017 Jul;12(4):441-447. doi: 10.1111/chd.12477. Epub 2017 May 19. PMID 28523732
- [Background] Reineke DC, Kaya A, Heinisch PP, Oezdemir B, Winkler B, Huber C, Heijmen RH, Morshuis W, Carrel TP, Englberger L. Long-term follow-up after implantation of the Shelhigh(R) No-React(R) complete biological aortic valved conduit. Eur J Cardiothorac Surg. 2016 Jul;50(1):98-104. doi: 10.1093/ejcts/ezv452. Epub 2015 Dec 30. PMID 26719402
- [Background] van den Berg J, de Bie S, Meijboom FJ, Hop WC, Pattynama PM, Bogers AJ, Helbing WA. Changes during exercise of ECG intervals related to increased risk for ventricular arrhythmia in repaired tetralogy of Fallot and their relationship to right ventricular size and function. Int J Cardiol. 2008 Mar 14;124(3):332-8. doi: 10.1016/j.ijcard.2007.02.009. Epub 2007 Apr 11. PMID 17433470
- [Background] Dallaire F, Wald RM, Marelli A. The Role of Cardiopulmonary Exercise Testing for Decision Making in Patients with Repaired Tetralogy of Fallot. Pediatr Cardiol. 2017 Aug;38(6):1097-1105. doi: 10.1007/s00246-017-1656-z. Epub 2017 Jun 16. PMID 28623384
- [Background] Schneider AW, Putter H, Klautz RJM, Bruggemans EF, Holman ER, Bokenkamp R, Hazekamp MG. Long-Term Follow-Up After the Ross Procedure: A Single Center 22-Year Experience. Ann Thorac Surg. 2017 Jun;103(6):1976-1983. doi: 10.1016/j.athoracsur.2016.11.064. Epub 2017 Feb 24. PMID 28242079